CLINICAL TRIAL: NCT03757026
Title: Balance Training Post Stroke: Intense Harnessed Multidirectional Training as Compared to Reactive and Conventional Protocols
Brief Title: Comparison of Three Balance Training Protocols for Individuals Post Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cleveland State University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, M. Ann Reinthal, Associate Professor, Cleveland State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2019-17; 18IPA34170316 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2018-11-13; First posted 2018-11-28 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Fall; Risk Reduction; Stroke; Balance
Keywords: Balance Training; Multidirectional harness; Conventional balance training; Reactive Slip Training; Stroke; Independent ambulation; Physical therapy
MeSH Terms: conditions — Risk Reduction Behavior; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physical Therapy (Active Comparator): 20-22 participants randomly assigned to receive 10 sessions of balance training. Conventional balance training group (PT) will receive individualized standard of care physical therapy with the goal of improving balance and mobility during sessions 3 through 12. The only instructions to the PT are that the focus of the course of care should be on "balance and mobility" and that there should be 10 sessions total. The first visit will include an initial evaluation and limited treatment. While the remaining 9 sessions will consist of 45 minutes of PT treatment.
  Interventions: Other: Conventional Physical Therapy
- Slip training (Experimental): 20-22 participants randomly assigned to 1 session of slip training and 9 sessions of accompanied walking. Reactive slip training group (Slip) will complete a standing slip session using the current protocol of scaling slip distance and force to each individual and modulating the slip intensity across the session based on subject responses. Initial perturbation intensity (percent body weight and slip distance) will be based on the participant's miniBEST score and each subsequent perturbation intensity will be determined based on their response to the previous perturbations. The remaining nine intervention sessions will consist of accompanied walking for up to 45 minutes. Participants will walk at a comfortable pace while accompanied by a researcher around Cleveland State.
  Interventions: Other: Slip Training
- Harnessed gaming (Experimental): 20-22 participants randomly assigned to 10 sessions of harnessed gaming. Multidirectional harness group (MHG) will use a harness with the multidirectional OASUS frame and play selected Kinect™ active video games with varied balance demands, while standing on multiple balance training surfaces (e.g., solid floor, rocker board, foam, slider platform). Participants will wear the fall-arresting harness in the OASUS system for all game play. Motion data will be collected during gaming for Sessions 2, 6, and 10. Each game/surface will be played for about 5 to 6 minutes for 4 game/surface conditions per session. All participants will progress with the prescribed sequence of games and surfaces, progressing based on their rating of the previous three bouts of play.
  Interventions: Other: Harnessed gaming

INTERVENTIONS:
Other: Conventional Physical Therapy — 20-22 participants randomly assigned to receive 10 sessions of balance training. Conventional balance training group (PT) will receive individualized standard of care physical therapy with the goal of improving balance and mobility during sessions 3 through 12. The only instructions to the PT are that the focus of the course of care should be on "balance and mobility" and that there should be 10 sessions total. The first visit will include an initial evaluation and limited treatment. While the remaining 9 sessions will consist of 45 minutes of PT treatment.
  Other Names: Balance training
  Arms: Conventional Physical Therapy
Other: Slip Training — 20-22 participants randomly assigned to 1 session of slip training and 9 sessions of accompanied walking. Reactive slip training group (Slip) will complete a standing slip session using the current protocol of scaling slip distance and force to each individual and modulating the slip intensity across the session based on subject responses. Initial perturbation intensity (percent body weight and slip distance) will be based on the participant's miniBEST score and each subsequent perturbation intensity will be determined based on their response to the previous perturbations. The remaining nine interventional sessions will consist of accompanied walking for up to 45 minutes. Participants will walk at a comfortable pace while accompanied by a researcher around Cleveland State.
  Other Names: Reactive slip training
  Arms: Slip training
Other: Harnessed gaming — 20-22 participants randomly assigned to 10 sessions of harnessed gaming. Multidirectional harness group (MHG) will use a harness with the multidirectional OASUS frame and play selected Kinect™ active video games with varied balance demands, while standing on multiple balance training surfaces (e.g., solid floor, rocker board, foam, slider platform). Participants will wear the fall-arresting harness in the OASUS system for all game play. Motion data will be collected during gaming for Sessions 2, 6, and 10. Each game/surface will be played for about 5 to 6 minutes for 4 game/surface conditions per session. All participants will progress with the prescribed sequence of games and surfaces, progressing based on their rating of the previous three bouts of play.
  Other Names: Multidirectional harness group
  Arms: Harnessed gaming

SUMMARY:
The purpose of this study is to compare conventional balance training to reactive training and to a novel, high intensity, harnessed training program. This study examines the impact of these interventions on fall risk and on a range of important aspects of balance including overall mobility, quality of life, and health. Participants will be 60-69 adults who had a stroke more than 6 months ago and who ambulate independently. Each participant will complete 14 sessions consisting of 4 (2 pre-, 2 post-) testing sessions and 10 intervention sessions. The pre and post testing will be the same and will consist of clinical and survey based balance and quality of life assessments and treadmill based perturbed gait testing.

The pretest will be sessions 1 and 2 will be followed by 10 intervention sessions. There will be 3 treatment groups: a conventional balance training group (PT), a reactive slip training group (Slip), and a multidirectional harness group (MHG). Participants will be randomly assigned to a group following screening and consent.

The conventional balance training group (PT) will receive 10 sessions of individualized standard of care physical therapy with the goal of improving balance and mobility. The only instructions to the PT are that the focus of the course of care should be on "balance and mobility" and that there should be 10 sessions.

The reactive slip training group (Slip) will complete a standing slip session using the current protocol of scaling slip distance and force to each individual and modulating the slip intensity across the session based on subject responses. The remaining nine intervention sessions will consist of accompanied walking for up to 45 minutes. Participants will walk at a comfortable pace while accompanied by a researcher.

The multidirectional harness group (MHG) will use a harness that allows movement in all directions, playing selected Kinect™ active video games with varied balance demands, on multiple balance training surfaces (e.g., rocker board, foam, slider platform). Participants will wear the fall-arresting harness for all game play. Motion data will be collected during Sessions 2, 6, and 10.

For all groups, two-post-test sessions will follow the intervention sessions and will be the same as the two-pretest session. The final session will also include reviewing the participants' falls diaries and setting up procedures for contacting participants weekly or biweekly about falls.

DETAILED DESCRIPTION:
This study compares conventional balance training to a reactive slip protocol and novel, high intensity, harnessed balance training using video gaming. It examines the impact of these three interventions on fall risk and on aspects of balance including overall mobility, quality of life and community participation. The study includes 60-69 adults who had a stroke more than 6 months ago and who walk independently. Participants will complete 14 sessions: 4 sessions (2 pre-, 2 post-) of testing and 10 intervention sessions. There will be one to two sessions per week depending on scheduling and participant preference.

The first session will begin with screening and the consent process after which participants will be randomly assigned to one of the following three groups of 20-22 participants each: conventional balance training (PT), reactive slip training (Slip), and multi-directional harnessed gaming training (MHG). The first individual entering the study will be randomly assigned to one of the three groups, the next person will be randomly assigned to one of the two remaining groups, and the third person will be placed in the remaining group. This process will be repeated with the next group of three individuals entering the study, and so on. Approximately midway through the study, researchers will assess group mix for impairment severity levels and adjust if necessary. All 14 sessions are outlined below including descriptions of testing and intervention procedures.

During session one, the screening, consent and randomization process will be followed by the clinical testing, falls history and falls diary initiation, then scheduling of subsequent visits. Participants will be questioned as to any falls within the last 12 months, and if any - how long ago for each fall and the circumstances of and any injuries from the fall as they recall them. The falls diary will be explained to the participants and participants will be asked to keep it during the weeks of the 14 sessions and for 6 months afterwards. The stability (RPS) scale will be explained to the participants and remaining clinical testing will be administered including the Mini-Balance Evaluation Systems Test (miniBEST). The limits of stability testing (LOS), including the reactive perturbation testing portion of the miniBEST will be performed with motion capture. If time, participant scheduling, and participant tolerance for activity permit, the LOS testing will be done at the second pre-test session because this will allow motion marker placement for one session rather than two, saving the participant time. If timing or participant activity tolerance do not allow, the LOS testing will be performed, with motion capture, at the first pre-test session.

The second session will continue the pre-test portion of the protocol with treadmill perturbation testing and LOS testing. All participants will be supported in a fall-arresting harness for all treadmill perturbation testing. First, the treadmill will be used to measure the participant's normal then fast walking speeds. For perturbations, the treadmill will be run at the participant's determined normal walking speed. It will randomly accelerate at mid-stance of the hemiparetic foot, then return to its usual speed. The participant will be asked to try to maintain his/her balance and continue walking as before, but that if the participant needs to stop, the investigator will halt the treadmill and provide a rest break. After each perturbation, the participant will be asked to score it on the RPS scale. Throughout all of the treadmill perturbation testing force, motion, and load cell data will be recorded and vital signs will be monitored consistent with Physical Therapy and exercise standards.

There will be up to 18 perturbations. The initial perturbation intensity will be based on the participant's miniBEST scores and normalized to that individual's maximum gait speed. Each subsequent perturbation intensity will be determined based on the participant's response to the previous perturbations: three consecutive falls (>30% of participant's body weight as measured by load cell) leads to a decrease in perturbation intensity; three consecutive recoveries (<5%of participant's body weight as measured by load cell) leads to an increase in perturbation intensity; and if the three previous perturbations were mixed (some combination of falls, recoveries, and harness assists) the perturbation will be unchanged. The outcome of each trial (fall, recovery, or harness assist) will be recorded.

After pretesting, 10 intervention sessions will begin based on group assignment, as described above. The conventional balance training group (PT) will receive individualized standard of care physical therapy with the goal of improving balance and mobility during sessions 3 through 12. This will be completed by an experienced community physical therapist who will be blinded to the other groups' activities and to all pre-testing results. The first visit will have approximately 60 minutes allotted for the initial evaluation and limited treatment while the remaining 9 sessions will consist of 45 minutes of PT treatment. The only instructions to the PT are that the focus of the course of care should be on "balance and mobility" and that there should be 10 sessions total. The investigators will be blinded to the specifics of the individual treatments provided by the PT(s).

The reactive slip training group (Slip) will complete one standing slip session using the current protocol of scaling slip distance and force to each individual and modulating the slip intensity across the session based on participant responses. To match intervention time to the other two groups, the remaining 9 sessions will involve 45 minutes of supervised walking with vital sign and distance monitoring, and rest as necessary.

All participants will use a full-body, fall-arresting harness throughout all slip testing. All participants will be informed that during the experimental procedures the Slip Trainer platform, on which they are standing, may move suddenly and unexpectedly under their feet. The participants will be asked to react as naturally as possible to the perturbation. The participants will also be informed that if they are unable to catch themselves, the full-body safety harness they will be wearing will prevent a fall from occurring. Participants will be reminded that they may request a rest break at any time. Participants will be guarded by an investigator (both licensed Physical Therapists) or by a Student PT supervised by an investigator.

The Slip Trainer is a low platform on rollers which allow only anterior-posterior (forward-backward) slips, not side to side. Participants will stand quietly on the trainer and slips will be induced by the (randomly timed and unannounced) release of weights from a designated height, causing the weights to fall and the platform to be pulled backward or forward approximately 15 - 30 centimeters. The amount of weight released will range from 15-40% of the participant's body weight. Up to 17 slips will be induced. The participants will self-rate their stability during the slip with the RPS immediately after each slip recovery. Motion, load cell and outcomes data will be collected throughout slip testing. Initial perturbation intensity (percent body weight and slip distance) will be based on the participant's miniBEST score and each subsequent perturbation intensity will be determined based on the participant's response to the previous perturbations. If this algorithm leads to the perturbations being reduced below 5% and 5 cm or above 40% and 30 cm, the trials will be stopped.

The remaining nine intervention sessions will consist of accompanied walking for up to 45 minutes. Participants will come to Cleveland State University and will walk at a comfortable pace while accompanied by a researcher in the areas in or adjacent to the Health Sciences spaces. Researchers will monitor the participants' vital signs as indicated and in the manner consistent with standard PT/exercise practice. Participants may request rest breaks as needed. The researcher will record the distances walked, the rests taken, and the vital signs as taken.

The multidirectional harness group (MHG) will use a harness with the Open Area Support System (OASUS) multidirectional harness framework and play selected Kinect™ active video games with varied balance demands, while standing on multiple balance training surfaces (e.g., solid floor, rocker board, foam, slider platform). Participants will wear the fall-arresting harness in the OASUS system for all game play. This harness allows participants to move freely in any direction except it limits their vertical descent to a pre-set height. This will be adjusted to a height that allows the participants to touch the floor or support surface with only their feet when fully suspended in the harness in any direction; no other body part will be able to reach the ground. This will be re-adjusted each time the participant changes the playing surface.

Initial game and training surface combinations as well as subsequent difficulty levels and training conditions will be chosen using a progression algorithm in conjunction with the Rate of Perceived Stability (RPS). Motion data will be collected during gaming for Sessions 2, 6, and 10. RPS scores will be collected during and immediately after all gaming sessions. Participants are able to use rest breaks and will be monitored throughout all sessions consistent with standard physical therapy/exercise practice. At the first session of MHG, participants will be introduced to each game and given time to practice playing that game until they feel comfortable with each game. All participants will progress with the prescribed sequence of games and surfaces, progressing based on their rating of the previous three bouts of play.

Two post-test sessions will follow the 10 intervention sessions. These will be equivalent to the two-pretest session above with the treadmill testing at session 13, LOS testing at either session 13 or 14, and the remaining clinical testing and follow up at session 14. All participants will be reminded of previous protocols/instructions completed in their pretest sessions. The 14th and final session will also include reviewing the participants' falls diaries and setting up procedures for contacting participants weekly or biweekly about falls. The participant will have a chance to ask any questions about the overall study and the payment forms will be signed.

ELIGIBILITY:
Inclusion Criteria:

* Stroke more than 6 months ago
* Self-identified balance issues
* Independent ambulation - specifically:

  * Walk at least one-half block (150') with or without standard cane or similar device
  * Stand independently for at least 30 seconds without physical assistance and without any device
  * At least ten steps without physical assistance and without any cane or similar device
* Ability to answer two-step questions

Exclusion Criteria:

* Allergic reaction to adhesive tapes
* Height above 74"
* Weight above 250 lbs
* Medical Condition - they are not eligible if they self-identify as having any musculoskeletal, neuromuscular, cardiopulmonary, or other conditions that would limit them from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Activities Specific Balance Confidence Scale (ABC) at study completion | Through study completion, on average three months.
  Indicates how self-confident the participants are not to lose their balance or become unsteady during specific activities like: walk around house, walk up and down stairs, pick up a slipper from the floor, etc. (Rating self-confidence from 0-100% on each of 16 items; then total score divided by 16 to give an overall self-confidence level, with 100% being fully confident on all 16 activities listed)
Change from baseline Mini Balance Evaluation Systems Test (MiniBEST) at study completion | Through study completion, on average three months.
  It aims to target and identify different balance control systems to identify balance deficits. The MiniBEST test is a 14-item test scored on a 3-level ordinal scale. Sections include anticipatory, reactive postural control, sensory orientation, and dynamic balance.
Change from baseline Mobility life space scale (MLSS) at study completion | Through study completion, on average three months.
  Questions for life-space mobility refers to 1) the level of the spatial area (bedroom, home, outside home, neighborhood, town, and beyond town) that an individual purposely moves through in daily life; 2) to the frequency of movement within a specific time in each area; and 3) the need for assistance with that movement. Scores range from 0 for someone who remains only the bedroom to up to 120 for someone who travels daily and independently out of his/her immediate community.
Change from baseline anterior, posterior, and lateral (to right and to left sides) limits of stability (LOS) scores at study completion | Through study completion, on average three months.
  Standing limits of stability (LOS) are tested by having the participant lean as far as he/she can to the front, back, and each side, twice, without stepping or needing to reach out for support. Motion data will be used to calculate the participant's center of mass (COM) and base of support (BOS) during this test. Then, the percent of the distance the participant can move his/her COM towards the edge of his/her BOS will be calculated in each of the four directions.
Change from baseline Treadmill perturbation stability scores at study completion | Through study completion, on average three months.
  Participants will walk on the treadmill to determine normal and maximum gait speed. Walking at normal speed, at a random time at about mid-stance of the hemiparetic lower extremity, the treadmill will accelerate suddenly then return to its previous speed. Initial perturbation intensity will be based on the participant's miniBEST scores and normalized to that individual's maximum gait speed. Each subsequent perturbation intensity will be based on the participant's response to previous perturbations: 3 consecutive falls (>30% of participant's body weight as measured by load cell) leads to a decrease in perturbation intensity; 3 consecutive recoveries (<5%) leads to an increase in perturbation intensity; and if the 3 previous perturbations were mixed (combination of falls, recoveries, and harness assists) the perturbation will be unchanged. Each response will be recorded as a recovery, harness assist, or fall (recovery <5%, harness assist 5%-30%, or fall >30% of body weight).
Change from baseline Falls Diary at 6 months post study completion | Through 6 months post study completion, on average a total of 9 months including study duration plus 6 months post study follow-up.
  During the pre-testing sessions, participants will be asked verbally to describe their recall of falls they have experienced in the past 12 months, to be recorded by a researcher, and to keep a log of falls over the course of the study and follow-up period of 6 months (to be collected monthly after end of study by phone call).

SECONDARY OUTCOMES:
Change from baseline Fugl Meyer Lower Extremity Sensory and Movement testing (FM LE) at study completion | Through study completion, on average three months.
  Evaluates and measures recovery in post-stroke hemiplegic patients. This outcome measure assesses sensorimotor function through the lower extremity. Items are scored on a 3-point ordinal scale.
Change from baseline Monofilament sensory testing (5.07 monofilament testing of foot and ankle) at study completion | Through study completion, on average three months.
  Using 5.07 monofilament, test the bottom and top of the foot below in locations pictured, including the medial and lateral malleolus and the anterior ankle at the mid-position between the two malleoli. While holding the handle, push the monofilament at a 90-degree angle against the skin until the monofilament bows. Hold for 1.5 seconds. Record with a check mark (√) if sensation intact and an X to denote no sensation at that point.
Change from baseline Five times sit-to-stand test (5XSTS) at study completion | Through study completion, on average three months.
  Patient sits with arms folded across chest and with back against the chair. With patients who have had a stroke, it is permissible to have the impaired arm at the side or in a sling.They must stand fully between repetitions of the test and not to touch the back of the chair during each repetition. They will stand up full 5 times. Documentation of speed and assist level (CGA, supervision, Mod I, or I) will be recorded.
Change from baseline Stroke Impact Scale (SIS) at study completion | Through study completion, on average three months.
  The Stroke Impact Scale (SIS) is a questionnaire that evaluates how a stroke has impacted the participant's health and life. The SIS has eight sections measuring self-perceived strength, memory and thinking, emotion, communication, activities of daily living, mobility, hand use, and work/leisure participation. There are multiple questions in each section, with each question rated from 1 to 5 in terms of activity difficulty, activity frequency, or strength. Summary scores are generated for each of the 8 sections. The scoring uses a transformed scale [(actual raw score - lowest possible raw score) /possible raw score range] x 100) and some items must be reverse scored. Scores range from 0-100% for each section with 100% indicating the highest level of function. There is also a final ninth section rating percent overall self-perceived recovery from the stroke with 100% being fully recovered.
Change from baseline Berg Balance Scale (BBS) at study completion | Through study completion, on average three months.
  The BBS measures balance ability (static and dynamic) among older adults. The BBS is a qualitative measure that assesses balance through performing functional activities. Each item is scored on a 5-point scale, ranging from 0 to 4, zero indicating the lowest level of function and 4 the highest level of function.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Reinthal, Principal Investigator — Cleveland State University
Locations (1):
- Cleveland State University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided